CLINICAL TRIAL: NCT00990691
Title: Pilot Study of the Effects of the Desipramine on the Neurovegetative Parameters of the Child With Rett Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-37; 2007-006739-30
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — Desipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desipramine high dose (Experimental): 12 patients with Rett syndrome receiving a daily dose of desipramine correlated with the weight :
  * From 15 to 25 kg : 50 mg ;
  * From 26 to 35 kg : 75 mg ;
  * From 36 to 45 kg : 100 mg ;
  * > 46 kg : 150 mg.
  Interventions: Drug: Administration of a high dose of desipramine
- Desipramine low dose (Experimental): 12 patients with Rett syndrome receiving a daily dose of desipramine correlated with the weight :
  * From 15 to 25 kg : 25 mg ;
  * From 26 to 35 kg : 50 mg ;
  * From 36 to 45 kg : 75 mg ;
  * > 46 kg : 100 mg.
  Interventions: Drug: Administration of a low dose of desipramine
- Placebo (Placebo Comparator): 12 patients with Rett syndrome receiving a daily dose of placebo.
  Interventions: Drug: Administration of a placebo

INTERVENTIONS:
Drug: Administration of a high dose of desipramine — Administration of a daily dose of desipramine correlated with the patient's weight :
  * From 15 to 25 kg : 50 mg ;
  * From 26 to 35 kg : 75 mg ;
  * From 36 to 45 kg : 100 mg ;
  * > 46 kg : 150 mg.
  Arms: Desipramine high dose
Drug: Administration of a low dose of desipramine — Administration of a daily dose of desipramine correlated with the patient's weight :
  * From 15 to 25 kg : 25 mg ;
  * From 26 to 35 kg : 50 mg ;
  * From 36 to 45 kg : 75 mg ;
  * > 46 kg : 100 mg.
  Arms: Desipramine low dose
Drug: Administration of a placebo — Administration of a daily dose of placebo
  Arms: Placebo

SUMMARY:
Rett syndrome is a neurodevelopmental disorder characterized by cognitive impairment, communication dysfunction, stereotypic movement disorder, and growth failure. Rett syndrome is caused by mutations in the Methyl CpG-Binding Protein-2 (MECP2) gene and has no treatment.

A mouse experimental model of Rett syndrome created by genetic invalidation of the MECP2 gene is available. It had been then observed that adult MECP2-deficient mice show respiratory alterations and found that endogenous noradrenaline helps to maintain a normal respiratory rhythm. Desipramine, a selective inhibitor of norepinephrine reuptake, seems to be efficient to reduce the respiratory alteration occuring in MECP2-deficient mice (Insem patent 2005, Villard and Roux 2006).

The aim of the study is to evaluate these obtained results in MECP2-deficient mice on patients with Rett syndrome.

DETAILED DESCRIPTION:
Rett syndrome is a neurodevelopmental disorder characterized by cognitive impairment, communication dysfunction, stereotypic movement disorder, and growth failure. The diagnosis of Rett syndrome is based on consensus clinical criteria. Rett syndrome is caused by mutations in the Methyl CpG-Binding Protein-2 (MECP2) gene and has no treatment.

Only a few improved cases have been reported concerning buspirone (Andaku, 2005, 1 patient), topiramate (Goyal, 2004, 8 patients), diazepam (Kurihara, 2001, 1 patient) and carnitin (Plochl, 2004, 1 patient).

Only one randomized study versus placebo has been published about a treatment by naltrexone including 25 patients. A light improvement of respiratory parameters was then observed with a deterioration of the cognitive function (Percy, 2004).

A mouse experimental model of Rett syndrome created by genetic invalidation of the MECP2 gene is available. It had been then observed that adult MECP2-deficient mice show respiratory alterations and found that endogenous noradrenaline helps to maintain a normal respiratory rhythm. Desipramine, a selective inhibitor of norepinephrine reuptake, seems to be efficient to reduce the respiratory alteration occuring in MECP2-deficient mice (Insem patent 2005, Villard and Roux 2006).

The aim of the study is to evaluate these obtained results in MECP2-deficient mice on patients with Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Rett syndrome;
* Girls weighing less than 60 kg;
* Respiratory alteration;
* Diagnosis of Rett syndrome confirmed by MECP2 genotyping (Xq28).

Exclusion Criteria:

* Boys;
* Pregnancy and breath feeding;
* Case history of status epilepticus;
* Patient treated by IMAO or sultopride;
* Hepatic or renal failure.

Ages: 4 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2014-08-11 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
To study the efficacy of the desipramine on the respiratory disturbations | 2 years

SECONDARY OUTCOMES:
To study the safety of the desipramine in the studied population | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Josette Mancini, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Mancini J, Dubus JC, Jouve E, Roux JC, Franco P, Lagrue E, Castelnau P, Cances C, Chaix Y, Rougeot-Jung C, Cornu C, Desportes V, Vallee L, Bahi-Buisson N, Truillet R, Attolini L, Villard L, Blin O, Micallef J. Effect of desipramine on patients with breathing disorders in RETT syndrome. Ann Clin Transl Neurol. 2017 Dec 27;5(2):118-127. doi: 10.1002/acn3.468. eCollection 2018 Feb. PMID 29468173